CLINICAL TRIAL: NCT00892099
Title: DIVINE: Dialysis Infection and Vitamin D In New England
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ravi Thadhani, Director of Clinical Research in Nephrology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009P-000398; R01DK084974 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal disease; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Dose Ergocalciferol (Experimental): Receives 50,000 IU of ergocalciferol weekly
  Interventions: Drug: Ergocalciferol
- Low Dose Ergocalciferol (Experimental): Receives 50,000 IU of ergocalciferol per month
  Interventions: Drug: Ergocalciferol
- Placebo (Placebo Comparator): Receives no ergocalciferol
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ergocalciferol — 50,000 IU tablet given weekly
  Other Names: vitamin D
  Arms: High Dose Ergocalciferol
Drug: Ergocalciferol — 50,000 IU tablet given monthly
  Other Names: Vitamin D
  Arms: Low Dose Ergocalciferol
Other: Placebo — Placebo equivalent of ergocalciferol, given weekly as one tablet
  Arms: Placebo

SUMMARY:
Infection is the second-leading cause of death in individuals requiring dialysis treatment for kidney failure. New research suggests the high risk of infection may be due in part to low levels of vitamin D, which are extremely common in kidney disease. This study is designed to determine safe and effective ways to raise vitamin D levels while monitoring effects on the immune system.

DETAILED DESCRIPTION:
We hypothesize that a profound deficiency of nutritional vitamin D (25-hydroxyvitamin D, 25D) in end-stage renal disease (ESRD) leads to an altered immune response, predisposing to early morbidity and mortality from infection, the second-leading cause of death in ESRD. In addition to impaired renal synthesis of the hormonal form of vitamin D (1,25-dihydroxyvitamin D; 1,25D), ESRD is accompanied by near universal insufficiency of 25D. In-vitro, ex-vivo, and retrospective human studies by our group and others suggest that 25D (and not 1,25D) is intimately linked to immune defense via alterations in the production of inflammatory cytokines and critical antimicrobial peptides including cathelicidin, which we have shown to identify ESRD subjects at risk for infection-related mortality. Ergocalciferol, which is rapidly converted to 25D, is the most widely available form of nutritional vitamin D in the US, yet guidelines to treat ESRD patients with nutritional vitamin D are absent because of limited data supporting its efficacy, safety, and biological effects in this population. To determine effective and safe doses of ergocalciferol in ESRD, we will perform a double blind placebo controlled randomized trial in 120 incident hemodialysis patients (40/arm x 3) with 25D levels < 30ng/ml, comparing two ergocalciferol dosing regimens (50,000 IU/week and 50,000 IU/month) and an identically appearing placebo. The primary outcome will be correction of vitamin D insufficiency (25D >30 ng/ml) at 12 weeks. Serum calcium and phosphate levels will be measured every 4 weeks to assess safety, and blood cytokine and cathelicidin levels will be measured every 4 weeks to determine biological responses. To examine biological effects in greater detail, a subset of subjects from each arm of the study will be further analyzed with serial macrophage gene expression profiles and whole blood cytokine profiles following ex-vivo stimulation with pro-inflammatory mediators (e.g., killed S. aureus). These experiments will inform us on how individuals with ESRD, based on their vitamin D status and the treatment they receive, may respond to infection. Laboratory measures will continue for 12 weeks. Clinical follow-up and monitoring for infection-associated events (including antibiotic use, rates of bacteremia, and sepsis) will continue for 20 weeks. This pilot trial addressing a significant unmet need in nephrology will involve basic, translational, and clinical investigators experienced in vitamin D research, infection and inflammation, and in trials involving ESRD subjects. These data will provide an important foundation for designing future clinical trials rigorously assessing the effect of nutritional vitamin D on infectious and other outcomes in ESRD.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Initiating chronic hemodialysis 3x/wk at Massachusetts General Hospital, Brigham and Women's Hospital or Beth Israel Deaconess Medical Center with planned transfer to Massachusetts chronic facility
* Serum 25D < 32 ng/ml
* Corrected serum calcium < 10.2 mg/dl
* Serum phosphate < 5.5 mg/dl
* Serum albumin > 3 g/dL
* Informed consent

Exclusion Criteria

* Pregnant or breastfeeding
* Women of childbearing potential not practicing one of the following measures of birth control: double-barrier method, hormonal contraceptives for at least 3 months prior to and during study, monogamous relationship with vasectomized partner, total abstinence from sexual intercourse with men during study.
* HIV positive
* History of allergic reaction to ergocalciferol
* Investigator considers subject unsuitable for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Thadhani, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Bhan I, Camargo CA Jr, Wenger J, Ricciardi C, Ye J, Borregaard N, Thadhani R. Circulating levels of 25-hydroxyvitamin D and human cathelicidin in healthy adults. J Allergy Clin Immunol. 2011 May;127(5):1302-4.e1. doi: 10.1016/j.jaci.2010.12.1097. Epub 2011 Feb 9. No abstract available. PMID 21310475
- [Result] Ishir Bhan, Dorothy A Dobens, Caitlin A. Trottier, Julia Beth Wenger, Hector Tamez, Joseph James Deferio, Kathryn J. Lucchesi, Ravi I. Thadhani. The DIVINE Trial: Dialysis Infection and Vitamin D in New England J. Am. Soc. Nephrol 24:2013 (Abstract: SA-PO1082)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Started | 36 | 33 | 36
Completed | 31 | 32 | 29
Not Completed | 5 | 1 | 7
Not completed — Death | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — replocated | 1 | 0 | 2
Not completed — Prolonged hospitalization | 1 | 0 | 1
Not completed — no further details | 1 | 0 | 1
Not completed — kidney function recovered | 0 | 1 | 0
Not completed — investigator decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo | Total
Number analyzed (Participants) | 36 | 33 | 36 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (17) | 58 (16) | 59 (17) | 57 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 7 | 23
  Male | 25 | 28 | 29 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 6 | 15
  Not Hispanic or Latino | 32 | 28 | 30 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 9 | 9 | 31
  White | 23 | 21 | 22 | 66
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
25(OH) vitamin D [Mean (Standard Deviation); unit: ng/ml] | 21.8 (7) | 22.3 (6.5) | 21.7 (7.3) | 21.9 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Serum 25D Level
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Number analyzed (Participants) | 36 | 33 | 36
ng/ml | 49.8 (2.3) | 38.3 (2.4) | 27.3 (2.3)

2. Secondary Outcome: Serum Calcium
Description: serum calcium levels (mg/dL)
Time Frame: every 4 weeks for 12 weeks
Population: Subject receiving treatment
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Number analyzed (Participants) | 36 | 33 | 36
mg/dl
  Visit 1 | 8.8 (0.1) | 8.7 (0.1) | 8.8 (0.1)
  Visit 2 | 9.1 (0.1) | 8.9 (0.1) | 9.0 (0.1)
  Visit 3 | 9.3 (0.1) | 9.1 (0.1) | 9.3 (0.1)
  Visit 4 | 9.1 (0.1) | 9.1 (0.1) | 9.1 (0.1)

3. Secondary Outcome: Serum Phosphate
Description: serum phosphate levels (mmol/L)
Time Frame: every 4 weeks for 12 weeks
Population: Subject receiving treatment
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Number analyzed (Participants) | 36 | 33 | 36
mmol/L
  Visit 1 | 4.2 (0.2) | 4.2 (0.2) | 4.1 (0.2)
  Visit 2 | 4.7 (0.3) | 4.7 (0.3) | 4.8 (0.3)
  Visit 3 | 4.9 (0.3) | 5.2 (0.3) | 5 (0.4)
  Visit 4 | 4.7 (0.3) | 5.4 (0.3) | 4.9 (0.3)

4. Secondary Outcome: Serum 25-OH Vitamin D
Description: serum 25-OH vitamin D levels (ng/mL)
Time Frame: every 4 weeks for 12 weeks
Population: Subject receiving treatment
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Number analyzed (Participants) | 36 | 33 | 36
ng/mL
  Visit 1 | 21.8 (1.2) | 21.7 (1.2) | 22.3 (1.2)
  Visit 2 | 42.2 (2.0) | 33.6 (2) | 27.6 (1.9)
  Visit 3 | 48.9 (2.2) | 35.6 (2.2) | 27 (2.1)
  Visit 4 | 49.8 (2.3) | 38.3 (2.4) | 27.4 (2.3)

5. Secondary Outcome: Serum 1,25(OH)2 Levels
Description: serum 1,25(OH) vitamin D levels (pg/mL)
Time Frame: At week 12
Population: Subject receiving treatment
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Number analyzed (Participants) | 36 | 33 | 36
pg/mL | 95 [66 to 135] | 100 [68 to 140] | 120 [62 to 149]

6. Secondary Outcome: Parathyroid Hormone
Description: serum PTH levels (pg/mL)
Time Frame: every 4 weeks for 12 weeks
Population: Subject receiving treatment
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Number analyzed (Participants) | 36 | 33 | 36
pg/mL
  Visit 1 | 281 (1) | 214 (1) | 243 (1)
  Visit 2 | 253 (1) | 195 (1) | 243 (1)
  Visit 3 | 255 (1) | 195 (1) | 196 (1)
  Visit 4 | 245 (1.1) | 216 (1) | 215 (1)

ADVERSE EVENTS:
Arm/Group | High Dose Ergocalciferol | Low Dose Ergocalciferol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 33/36 | 26/33 | 28/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Ergocalciferol (N=36) | Low Dose Ergocalciferol (N=33) | Placebo (N=36)
Elevated phosphorus (Renal and urinary disorders) | 13 (13) | 13 (13) | 15 (15)
Elevated calcium (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Elevated PTH (Endocrine disorders) | 6 (6) | 2 (2) | 4 (4)
Elevated potassium (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Elevated white blood count (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Low albumin (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization (Surgical and medical procedures) | 14 (14) | 11 (11) | 13 (13)
Infection (Infections and infestations) | 11 (11) | 11 (11) | 8 (8)
Cardiovascular (Cardiac disorders) | 6 (6) | 2 (2) | 3 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Fluid overload (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea/vomiting/diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3)
Hypotension (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1)
Other (General disorders) | 4 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No